CLINICAL TRIAL: NCT01261598
Title: Predictive Value of FDG-TEP During Radiotherapy (RT) or Chemo-radiotherapy (CRT) in Patients With Non Small Cell Lung Cancer on the One-year Survival
Brief Title: Predictive Value of FDG-TEP During Radiotherapy or Chemo-radiotherapy in Patients With NCSC on the One-year Survival
Acronym: RTEP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHB06-02
Record Dates: First submitted 2010-11-19; First posted 2010-12-16 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer; NSCLC
Keywords: Positron-Emission Tomography; PET Scan; Non-Small-Cell Lung Carcinoma; Radiation Oncology; SUV
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Patients treated with curative and exclusive radiotherapy (60 Gy minimum), with possibly prior chemotherapy
  Interventions: Procedure: Positron Emission Tomography
- 2 (Other): Patient treated with concomitant chemotherapy and radiotherapy (60 Gy minimum), with possibly prior chemotherapy chemotherapy Treatment
  Interventions: Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Positron Emission Tomography — Positron Emission Tomography
  Other Names: PET scan

SUMMARY:
The poor prognosis in the early-stage of lung cancer is due to potential worsening of the disease (local relapse, metastasis), to insufficient efficacy and toxicity of actual treatments.

FDG-PET is a medical imaging modality allowing the quantification of the tumour glucose consumption. Then, this exam is used for pathology staging, target volume definition for RT, and treatment efficiency few months after RT or CRT. Our assumption is that an FDG-PET exam during the course of the RT or CRT might be predictive of the treatment efficiency few months later.

In this study, the investigators propose to perform 4 FDG-PET: first "PET1" before radiotherapy, second "PET2" during the radiotherapy (see RTEP1), third and fourth "PET3" "PET4" 3month and 12 month after the therapy.

The investigators will investigate the performances of FDG-PET performed during the RT or CRT for the prediction of the one-year patient heath outcome. If the predictive value of TEP2 is confirmed, the investigators would be able to optimize the planning treatment during the course of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* Fertile patients must use effective contraception
* WHO performance status <2
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (≥ 10 mm with spiral CT scan)

Exclusion Criteria:

* Pregnant or lactating females
* Baseline fludeoxyglucose F 18 (FDG)-positron emission tomography (PET) scan without any target lesion
* Unable to under PET CT evaluation
* other concurrent investigational agents
* No Planning to undergo curative intent radiotherapy
* familial, social, geographic, or psychological conditions that would preclude study participation
* Prior malignancy progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
SUV max from FDG PETScan | Baseline - 5 Weeks after begining of radiotherapy- 3 months after end of radiotherapy- 1 year afterwards
  Measure of FDG-TEP uptake variation (SUV max) to assess predictive value of FDG-TEP during radiotherapy

SECONDARY OUTCOMES:
Study of several optimized radiotherapy scenary according to the quantification of the tumour glucose consumption during radiotherapy | after the completion enrollment date

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DUBRAY, phD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganem J, Thureau S, Gardin I, Modzelewski R, Hapdey S, Vera P. Delineation of lung cancer with FDG PET/CT during radiation therapy. Radiat Oncol. 2018 Nov 12;13(1):219. doi: 10.1186/s13014-018-1163-2. PMID 30419929
- [Derived] Calais J, Thureau S, Dubray B, Modzelewski R, Thiberville L, Gardin I, Vera P. Areas of high 18F-FDG uptake on preradiotherapy PET/CT identify preferential sites of local relapse after chemoradiotherapy for non-small cell lung cancer. J Nucl Med. 2015 Feb;56(2):196-203. doi: 10.2967/jnumed.114.144253. Epub 2015 Jan 8. PMID 25572091
- [Derived] Vera P, Mezzani-Saillard S, Edet-Sanson A, Menard JF, Modzelewski R, Thureau S, Meyer ME, Jalali K, Bardet S, Lerouge D, Houzard C, Mornex F, Olivier P, Faure G, Rousseau C, Mahe MA, Gomez P, Brenot-Rossi I, Salem N, Dubray B. FDG PET during radiochemotherapy is predictive of outcome at 1 year in non-small-cell lung cancer patients: a prospective multicentre study (RTEP2). Eur J Nucl Med Mol Imaging. 2014 Jun;41(6):1057-65. doi: 10.1007/s00259-014-2687-9. Epub 2014 Feb 22. PMID 24562641